CLINICAL TRIAL: NCT01760018
Title: Comparison Between Propofol-remifentanil Total Intravenous Anesthesia and Desflurane-remifentanil Balanced Anesthesia With Regard to Post-anesthetic Functional Recovery Measured With QoR-40
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 4-2012-0748
Record Dates: First submitted 2012-12-31; First posted 2013-01-03 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Thyroid Operation Under General Anesthesia
Keywords: desflurane, total intravenous anesthesia, QoR-40

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desflurane group (Experimental)
  Interventions: Drug: desflurane group
- TIVA(total intravenous anesthesia) group (Active Comparator)
  Interventions: Drug: TIVA group

INTERVENTIONS:
Drug: desflurane group — anesthesia is maintained with desflurane and remifentanil (Desflurane group)
  Arms: Desflurane group
Drug: TIVA group — anesthesia is maintained with fresofol and remifentanil (TIVA group).
  Arms: TIVA(total intravenous anesthesia) group

SUMMARY:
Total intravenous anesthesia (TIVA) and inhalation anesthesia are both widely and safely used, and there are many clinical trials comparing these on various aspects of anesthesia. However, there have not been studies comparing the quality of recovery from the different methods of general anesthesia. In this study, the investigators compare the functional recovery after general anesthesia in TIVA and inhalation anesthesia with QoR-40 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* patients who are undergoing thyroid operation belong to ASA class 1 or 2

Exclusion Criteria:

* patients who are belongs to ASA class 3 or more,
* patients who have underlying complicated cardiovascular or psychological disease.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
QoR-40 score | at 24 hours later after surgery
  QoR-40 score is going to be measured at preoperative period, 24 hours, and 48 hours later after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540
- [Derived] Lee WK, Kim MS, Kang SW, Kim S, Lee JR. Type of anaesthesia and patient quality of recovery: a randomized trial comparing propofol-remifentanil total i.v. anaesthesia with desflurane anaesthesia. Br J Anaesth. 2015 Apr;114(4):663-8. doi: 10.1093/bja/aeu405. Epub 2014 Dec 10. PMID 25500679